CLINICAL TRIAL: NCT01120561
Title: An Expanded Access, Open-Label Study of Trastuzumab-MCC-DM1 Administered Intravenously to Patients With HER2- Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Trastuzumab-MCC-DM1 in Patients With HER2- Positive Locally Advanced or Metastatic Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TDM4884g
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
Keywords: TDM-1 EAP; T-DM1 EAP; TDM1 EAP; Trastuzumab-MCC-DM1 EAP; Trastuzumab emtansine; EAP; T-PAS
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

INTERVENTIONS:
Drug: trastuzumab-MCC-DM1 — Intravenous repeating dose

SUMMARY:
This is a multicenter, open-label, single-arm, expanded access study designed to provide T-DM1 to patients with HER2-positive locally advanced or metastatic breast cancer and to evaluate the safety and efficacy of T-DM1 administered by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented breast cancer
* Locally advanced or metastatic breast cancer
* HER2-positive breast cancer documented as FISH-positive, IHC 3 + or CISH-positive by local laboratory assessment
* Histologically or cytologically confirmed invasive breast cancer: incurable, unresectable, locally advanced breast cancer previously treated with multimodality therapy or metastatic breast cancer
* Prior treatment for breast cancer in the adjuvant, unresectable, locally advanced, or metastatic setting must include both: a taxane, alone or in combination with another agent, and Trastuzumab, alone or in combination with another agent in the adjuvant, unresectable, locally advanced, or metastatic setting
* Documented progression of incurable unresectable, locally advanced, or metastatic breast cancer during their most recent treatment regimen
* Progression must occur during or after most recent treatment for locally advanced/metastatic breast cancer or within 6 months after completing adjuvant therapy
* Adequate hematologic and end organ function
* Agreement to use an effective form of birth control throughout the study
* Life expectancy ≥ 90 days as assessed by the investigator

Exclusion Criteria:

* Less than 14 days from the first study treatment since the last anti-cancer therapy, including chemotherapy, biologic, experimental, immune, hormonal or endocrine therapy
* Prior T-DM1 therapy
* History of exposure to cumulative doses of select anthracyclines
* History of intolerance or hypersensitivity to trastuzumab, murine proteins, or any of the excipients, that resulted in trastuzumab being permanently discontinued
* Brain metastases that are untreated or progressive or currently require any type of therapy, including radiation, surgery, and/or steroids to control symptoms from brain metastases within 30 days before the first study treatment
* Peripheral neuropathy of Grade ≥ 3 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0, at the time of the first study treatment
* History of clinically significant cardiac dysfunction
* Current known active infection with HIV, hepatitis B virus, or hepatitis C virus
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to first study treatment
* Pregnancy or lactation

NOTE: The site selection process has been completed. Patients can enroll at participating sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-05

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (15):
- United States (15):
  - Investigational Site, Highland, California
  - Investigational Site, Stockton, California
  - Investigational Site, Denver, Colorado
  - Investigational Site, Plantation, Florida
  - Investigational Site, Lafayette, Indiana
  - Investigational Site, Cedar Rapids, Iowa
  - Investigational Site, Scarborough, Maine
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Clarkson Valley, Missouri
  - Investigational Site, Farmington, New Mexico
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Charleston, South Carolina
  - Investigational Site, Fairfax, Virginia
  - Investigational Site, Seattle, Washington